CLINICAL TRIAL: NCT00764504
Title: Encore Reverse Shoulder Prosthesis
Brief Title: Reverse Shoulder Prosthesis Study
Acronym: RSP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Encore Medical, L.P. (Industry)
Responsible Party: Jane M. Jacob Ph.D., DJO Surgical
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Study 300
Record Dates: First submitted 2008-09-30; First posted 2008-10-02 (Estimated); Results first posted 2011-04-19 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-03

CONDITIONS: Rotator Cuff Arthropathy; Failed Total Shoulder; Failed Hemi-arthroplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Primary (Experimental): Primary shoulder
  Interventions: Device: Reverse Shoulder Prosthesis
- Revision (Experimental): Revision shoulder
  Interventions: Device: Reverse Shoulder Prosthesis
- Continued Access (Experimental): Primary shoulder subjects enrolled at a later date in order to collect more data.
  Interventions: Device: Reverse Shoulder Prosthesis

INTERVENTIONS:
Device: Reverse Shoulder Prosthesis — For subjects with rotator cuff arthropathy and no previous shoulder device implanted.
  Arms: Continued Access; Primary
Device: Reverse Shoulder Prosthesis — For subjects with rotator cuff arthropathy and a failed hemi or total shoulder implant.
  Arms: Revision

SUMMARY:
The objective of this clinical study is to evaluate the safety and efficacy of the Encore Reverse Shoulder Prosthesis (RSP). The clinical results of the RSP will be compared to clinical results published in literature for rotator cuff arthropathy and salvage procedures.

ELIGIBILITY:
Inclusion Criteria:

* Irreparable rotator cuff or failed hemi or total shoulder arthroplasty with irreparable rotator cuff
* Evidence of upward displacement of the humeral head with respect to the glenoid
* Loss of glenohumeral joint space
* Functional deltoid muscle
* Patient is likely to be available for evaluation for the duration of the study
* Visual Analog Pain Scale 5 or greater

Exclusion Criteria:

* Non functional deltoid muscle
* Active sepsis
* Excessive glenoid bone loss
* Pregnancy
* Neurological abnormalities, which could hinder patient's ability or willingness to follow study procedures. For example, any that may restrict physical activities such as Parkinson's, Multiple Sclerosis, or previous stroke, which affects upper extremity.
* Mental conditions that may interfere with ability to give an informed consent or willingness to fulfill the study requirements (i.e., severe mental retardation such that the patient cannot understand the informed consent process, global dementia, prior strokes that interfere with the patient's cognitive abilities, senile dementia, and Alzheimer's Disease.
* Prisoners
* Conditions that place excessive demand on the implant (i.e. Charcot's joints, muscle deficiencies, refusal to modify postoperative physical activities, skeletal immaturity).
* Known metal allergy (i.e., jewelry).
* Visual Analog Pain Scale <5.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 516 (Actual)
Dates: Start 2002-10; Primary Completion 2008-06 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Frankle, M.D., Principal Investigator — Florida Orthopedic Institute
Locations (25):
- United States (25):
  - Arthritis Orthopedics and Sports Medicine, Glendale, California
  - Orthopaedic Specialty Institute, Orange, California
  - University of Colorado, Denver, Colorado
  - Orthopedic Center of the Rockies, Fort Collins, Colorado
  - Advanced Orthopedic and Sports Medicine Specialists, P.C., Lonetree, Colorado
  - Steadman Hawkins SPT Medical Foundation, Vail, Colorado
  - Atlantis Orthopaedics, Atlantis, Florida
  - Orthopaedic Surgery & Sports Medicine, Jupiter, Florida
  - Palm Beach Orthopaedic Institute, Palm Beach Gardens, Florida
  - Florida Orthopedic Institute, Temple Terrace, Florida
  - Atlanta, Georgia
  - Cincinnati Sports Medicine & Orthopaedic Center, Crestview, Kentucky
  - Lutherville, Maryland
  - Orthopedic Specialists, Towson, Maryland
  - TRIA Orthopaedic Center, Bloomington, Minnesota
  - Hospital for Special Surgery, New York, New York
  - UNC School of Medicine, Chapel Hill, North Carolina
  - Crystal Clinic, Akron, Ohio
  - Bone & Joint Hospital, LLC, Oklahoma City, Oklahoma
  - Orthopedic Research Foundation of the Carolinas, Spartanburg, South Carolina
  - The Carrell Clinic, Dallas, Texas
  - Orthopedic Associates of Dallas, Dallas, Texas
  - Orthopedic Specialty Associates, P.A., Fort Worth, Texas
  - Unlimited Research, San Antonio, Texas
  - Orthopedic Institute, Tyler, Texas

REFERENCES:
- See also: Sponsor company home page — http://www.djosurgical.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Primary: Subjects who are eligible to receive a reverse shoulder prosthesis and who have not previously received another orthopedic implant in the operative shoulder.
- Revision: Subjects who are eligible to receive a reverse shoulder prosthesis and who have previously received another orthopedic implant in the operative shoulder. The change in implant device is due to failure of the previously inserted orthopedic device.
- Continued Access: Subjects who are eligible to receive a reverse shoulder prosthesis and who have not previously received another orthopedic implant in the operative shoulder. This group are also primary subjects who were enrolled at a later date in order to collect additional data on the reverse shoulder.
Period: Overall Study
Arm/Group | Primary | Revision | Continued Access
Started | 141 | 141 | 234
Completed | 75 | 71 | 131
Not Completed | 66 | 70 | 103
Not completed — Death | 12 | 6 | 13
Not completed — Revision of Device | 12 | 23 | 14
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 7 | 4
Not completed — Lost to Follow-up | 40 | 34 | 72

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Primary | Revision | Continued Access | Total
Number analyzed (Participants) | 141 | 141 | 234 | 516
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 30 | 52 | 57 | 139
  >=65 years | 111 | 89 | 177 | 377
Age Continuous [Mean (Standard Deviation); unit: years] | 71.9 (9.5) | 67.4 (11.6) | 71.2 (9.2) | 70.4 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 97 | 136 | 320
  Male | 54 | 44 | 98 | 196
Region of Enrollment [Number; unit: participants]
  United States | 141 | 141 | 234 | 516
Operative Shoulder [Number; unit: participants]
  Right | 87 | 83 | 146 | 316
  Left | 54 | 58 | 88 | 200

OUTCOME MEASURES:

1. Primary Outcome: American Shoulder and Elbow Surgeons Shoulder Score
Description: The patient self-report section of the ASES is a condition specific scale which is intended to measure functional limitations and pain of the shoulder. On a scale of 0 to 100, the use of their shoulder is measured with 0 = no use and 100 = full use. The assessment is done in two sections. One Pain (measured by the Visual Analog Pain Scale) and the second is a list of 10 questions referred to as the Activities of Daily Living. The results are calculated with the following equation:
  [(10 - Visual analog scale pain score) x 5] + [(5/3) x Cumulative ADL score]
Time Frame: 2-year
Population: The number of participants analyzed is based on the number of participants who completed the study at the 2 year time frame and who had complete data sets at the final visit.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Primary | Revision | Continued Access
Number analyzed (Participants) | 59 | 49 | 98
Units on a scale | 76 (18.5) | 62 (18.5) | 77 (18.1)

2. Primary Outcome: Average Range of Motion
Description: Physician's assessment of a subject's range of motion in degrees.
Time Frame: 2-year
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Angle of Degrees of Shoulder Motion
Arm/Group | Primary | Revision | Continued Access
Number analyzed (Participants) | 59 | 49 | 98
Angle of Degrees of Shoulder Motion
  Active forward elevation | 119.6 (39.3) | 84.4 (36.5) | 120.4 (34.7)
  Active external rotation | 33.3 (19.0) | 23.3 (18.7) | 37.1 (24.2)
  Active cross body adduction | 25.8 (18.6) | 13.9 (15.6) | 27.4 (20.6)

3. Primary Outcome: Subject Satisfaction With Surgery
Description: Each subject had a chance to rate their satisfaction with surgery at each study interval.
Time Frame: 2-year
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Primary | Revision | Continued Access
Number analyzed (Participants) | 59 | 49 | 98
participants
  Excellent | 31 | 20 | 60
  Good | 18 | 12 | 27
  Satisfactory | 6 | 13 | 9
  Unsatisfactory | 4 | 4 | 2

4. Primary Outcome: Have Surgery Again?
Description: Subject satisfaction: subject's willingness to have surgery performed again if necessary.
Time Frame: 2-year
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Primary | Revision | Continued Access
Number analyzed (Participants) | 59 | 49 | 98
participants
  Yes | 52 | 40 | 88
  No | 7 | 9 | 10

5. Primary Outcome: Neer's "Limited Goals"
Description: To meet Neer's limited goals, a subject must report: none, slight or moderate pain with unusual activity and exhibit >90 degrees active forward elevation and exhibit >20 degrees of active external rotation.
Time Frame: 2-year
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Primary | Revision | Continued Access
Number analyzed (Participants) | 59 | 49 | 98
participants
  Yes - criteria met | 33 | 9 | 59
  No - criteria not met | 26 | 40 | 39

6. Primary Outcome: Radiographic Failures
Description: Radiographic failure is defined as a shift in the position of the component >3mm or 3 degrees, a fracture of the cement mantle, a fracture of the component, or a >2mm radiolucency completely around either prosthesis.
Time Frame: Post-operative, 3-month, 6-month, 1-year, 2-year
Population: Number of subjects who came in for a 2 year visit and completed the x-ray portion of the exam.
Measure: Number; unit: participants
Arm/Group | Primary | Revision | Continued Access
Number analyzed (Participants) | 69 | 62 | 127
participants | 0 | 0 | 0

7. Primary Outcome: Safety Assessment
Description: Number of device related adverse events and device failures at the 2 year time frame.
Time Frame: 2-year
Population: Adverse events were collected for all subjects who received the RSP device whether or not they were removed from the study at a later date due to protocol violation or consent issues.
Measure: Number; unit: adverse events
Arm/Group | Primary | Revision | Continued Access
Number analyzed (Participants) | 156 | 162 | 249
adverse events
  Revisions of device | 12 | 23 | 14
  Number of device related adverse events | 27 | 25 | 14
  Total number of operative site adverse events | 87 | 117 | 91

ADVERSE EVENTS:
Arm/Group | Primary | Revision | Continued Access
Serious Adverse Events (participants affected / at risk) | 0/156 | 0/162 | 0/249
Other Adverse Events (participants affected / at risk) | 116/156 | 113/162 | 157/249
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primary (N=156) | Revision (N=162) | Continued Access (N=249)
Anemia / Bleeding (Blood and lymphatic system disorders) | 1 (1) | 8 (9) | 0 (0)
Broken Device / Component (Surgical and medical procedures) | 4 (4) | 2 (2) | 0 (0)
Broken Screw (Surgical and medical procedures) | 9 (11) | 3 (3) | 2 (2) — screws are used to secure parts of the device to bone and will occasionally break.
Cancer (Immune system disorders) | 5 (5) | 3 (3) | 5 (5)
Death - Natural Causes (Social circumstances) | 9 (9) | 5 (5) | 13 (13)
Device Instability / Failure (Surgical and medical procedures) | 11 (11) | 16 (17) | 8 (8) — Device became unstable or failed which required a revision surgery.
Dislocation (Musculoskeletal and connective tissue disorders) | 9 (14) | 21 (25) | 9 (13)
Edema (Blood and lymphatic system disorders) | 5 (5) | 7 (8) | 4 (4)
Fracture (Musculoskeletal and connective tissue disorders) | 16 (16) | 16 (16) | 21 (23)
Heart Complications (Cardiac disorders) | 10 (11) | 3 (5) | 11 (11)
Infections (Infections and infestations) | 4 (4) | 13 (18) | 16 (17)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 57 (81) | 47 (64) | 68 (103)
Neurological disorder and numbness (Nervous system disorders) | 4 (4) | 5 (5) | 8 (8)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 7 (7)
Stroke (Vascular disorders) | 2 (2) | 1 (1) | 4 (6)
Swelling (Vascular disorders) | 3 (3) | 3 (3) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less